CLINICAL TRIAL: NCT04253574
Title: Comparison of 18F-2-fluoro-2-deoxy-D-glucose (18F-FDG) PET/CT and Ultrasound in Staging of Patients With Malignant Melanoma: An Analysis in a Single Patient Population
Brief Title: Comparison of PET/CT and Ultrasound in Staging of Malignant Melanoma
Status: Completed | Type: Observational
Sponsor: University of Basel (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Joachim Hohmann, Associate Professor, University of Basel
Other Study IDs: UBaselMM
Record Dates: First submitted 2020-01-26; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Malignant Melanoma
Keywords: Malignant Melanoma; Staging; 18F-FDG PET/CT; Ultrasound
MeSH Terms: conditions — Melanoma | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with malignant melanoma: 258 patients (w: 112, m: 146 age: 61±16 years) met the primary inclusion criteria. They were all examined by 18F-FDG PET/CT, 176 patients additionally by US (peripheral lymph nodes (pUS) and/or abdomen (aUS)).
  Interventions: Diagnostic Test: Imaging with 18F-FDG PET/CT and/or Ultrasound

INTERVENTIONS:
Diagnostic Test: Imaging with 18F-FDG PET/CT and/or Ultrasound — All patients were all examined by 18F-FDG PET/CT, 176 patients additionally by US (peripheral lymph nodes (pUS) and/or abdomen (aUS)) in the search of primary tumors or metastases of their malignant melanomas.

SUMMARY:
This is the first study which evaluates the different staging modalities 18F-2-fluoro-2-deoxy-D-glucose PET/CT (PET/CT) and diagnostic ultrasound (US) in a single patient cohort with malignant melanoma (MM). Previous analyses are ambivalent regarding the modality of choice. These analyses, however, compared separate patient cohorts for each modality.

Inclusion criteria were a primary staging or re-staging of suspected or confirmed MM with one or more PET/CT and/or one or more US. Exclusion criteria were the non-existence of a malignancy or a malignancy other than MM, alone or in combination with an MM.

The analysis includes the calculation of sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy in a per-patient (PPA), per-examination (PEA) and per-lesion analysis (PLA). This was done individually for PET/CT and US, and in PLA also for the combination of these two radiological modalities. Furthermore, US was divided into US as a whole (wUS), peripheral lymph nodes (pUS) and/or abdomen (aUS).

The principle equivalence of the two imaging modalities is set up as a null hypothesis H0 in all three analyses. As a further null hypothesis H0, the equivalence of the combined application compared to the sole applications of the two imaging modalities is asserted. The aim is the refutation of the null hypothesis H0 by significant differences in sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* the existence of malignant melanoma (MM) as primary tumour or metastases

Exclusion Criteria:

* the non-existence of a malignancy,
* a malignancy other than MM, alone or in combination with an MM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 258 patients (112 (43%) women, 146 (57%) men, mean age: 61 ± 16 years)
  Melanoma subtypes:
  * nodular subtype (n = 68, 35% of the classified melanomas)
  * superficial-spreading subtype (n = 61, 32%)
  * acral lentiginous melanoma (n = 12, 6%)
  * lentigo maligna (n = 7, 4%)
  * rare subtypes (n = 44, 23%)
  * melanoma without characterisation (n = 66)
  At first diagnosis:
  * 224 patients (87%) with a primary tumor only
  * 34 patients (13%) with metastases only
  Location of the melanoma lesion:
  * head or neck: 48 patients
  * trunk: 102 patients
  * upper limbs: 42 patients
  * lower limbs: 66 patients
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of 18F-FDG PET/CT and ultrasound regarding the detection of primary tumours and metastases of melanoma | September 1998 - August 2014
  The principle equivalence of the two imaging modalities is set up as a null hypothesis H0 in a per-patient (PPA), per-examination (PEA) and per-lesion analysis (PLA). As a further null hypothesis H0, the equivalence of the combined application compared to the sole applications of the two imaging modalities is asserted. The aim is the refutation of the null hypothesis H0 by significant differences in sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Hohmann, MD MSc, Principal Investigator — University of Basel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xing Y, Bronstein Y, Ross MI, Askew RL, Lee JE, Gershenwald JE, Royal R, Cormier JN. Contemporary diagnostic imaging modalities for the staging and surveillance of melanoma patients: a meta-analysis. J Natl Cancer Inst. 2011 Jan 19;103(2):129-42. doi: 10.1093/jnci/djq455. Epub 2010 Nov 16. PMID 21081714
- See also: Independent Institute for Quality and Efficiency in Health Care (IQWiG) final report on MM staging [German] — https://www.iqwig.de/download/D06-01F_Abschlussbericht_PET_und_PET-CT_bei_malignem_Melanom.pdf